CLINICAL TRIAL: NCT02011191
Title: Biotin Deficiency and Restless Legs Syndrome: Evidence for a Causal Relationship From Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Biotin Deficiency and Restless Legs Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidi Moretti, MS, RD (Other)
Collaborators: Saint Patrick Hospital (Other); University of Arkansas (Other)
Responsible Party: Sponsor-Investigator, Heidi Moretti, MS, RD, Clinical Dietitian, Saint Patrick Hospital
Organization: Saint Patrick Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NIH DK 36823-28
Record Dates: First submitted 2012-01-03; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: End Stage Renal Disease; Restless Legs Syndrome
Keywords: Biotin; Restless; Kidney; Dialysis; Renal
MeSH Terms: conditions — Kidney Failure, Chronic; Restless Legs Syndrome; Psychomotor Agitation | interventions — Biotin; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biotin (Active Comparator): 10,000 micrograms biotin daily for 8 weeks
  Interventions: Dietary Supplement: Biotin Supplementation
- Sugar pill (Placebo Comparator)
  Interventions: Dietary Supplement: Sugar Pill

INTERVENTIONS:
Dietary Supplement: Biotin Supplementation — 10,000 micrograms biotin supplement daily for 8 weeks
  Other Names: Biotin, Hillestad Pharmeceuticals
  Arms: Biotin
Dietary Supplement: Sugar Pill — Identical sugar pill, identical bottle as the biotin supplementation group
  Other Names: Hillestad Pharmeceuticals
  Arms: Sugar pill

SUMMARY:
Restless Leg Syndrome (RLS) is a common neuropathic disorder in patients with end stage renal disease (ESRD). Study Design: Because micronutrient depletion has been associated with RLS in ESRD and because the vitamin biotin is dialyzable, the investigators examined the relationship between biotin status and RLS in ESRD. Objectives: To assess the prevalence of biotin deficiency in those with and without RLS (Study 1) and to determine the effect of biotin supplementation on RLS symptoms (Study 2) in patients receiving chronic dialysis due to ESRD.

DETAILED DESCRIPTION:
Setting and Participants: ESRD patients receiving chronic dialysis as outpatients at Saint Patrick Hospital in Missoula, Montana.

ELIGIBILITY:
Inclusion Criteria:

* ESRD requiring hemodialysis or peritoneal dialysis therapy for a duration of at least 3 months.

Exclusion Criteria:

* History of consumption of more than 300 micrograms daily of biotin
* Oral contraceptive therapy containing high amounts of estrogen because studies in rats provide evidence that high doses of steroid hormones reduce biotin status {Wang, 1997 #1634}
* Women of childbearing age because of concern that biotin deficiency may be teratogenic {Mock, 2009 #2568}.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Biotin Status of Dialysis Patients | Measurement at baseline and after 8 weeks of treatment
  Biotin status is measured using Propionyl CoA carboxylase and Propionyl CoA carboxylase activation coefficients that are from isolated lymphocyte samples. This is a measurement that is independent of kidney function.
Change in Restless Legs Syndrome (RLS) symptoms after Biotin treatment | Baseline RLS score measurement and measurement after 8 weeks of treatment
  The RLS is measured using the International Restless Legs Syndrome Scale, a validated tool for assessing severity of RLS in patient who have been diagnosed with RLS.

CONTACTS AND LOCATIONS:
Overall Officials: John Lakatua, MD, Principal Investigator — Saint Patrick Hospital